CLINICAL TRIAL: NCT04388319
Title: Zonisamide/Bupropion Effects on Switching to Electronic Cigarettes
Acronym: BuZonE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BuZonE
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Smoking Cessation
Keywords: e-cigarette; zonisamide; bupropion; combustible cigarettes
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Zonisamide; Bupropion; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination zonisamide and bupropion with e-cigarette (Experimental): Participants enrolled in the study will receive a G6 e-cigarette at V2 for ad libitum use. After the first week of e-cigarette use, (at V3) participants will be given zonisamide and bupropion in addition to continued use of the G6. Use of these study drugs will continue for 12- weeks with a target complete switch date (from combustible cigarettes to e-cigarettes) one week after study drug initiation.
  Interventions: Drug: Zonisamide; Drug: Bupropion; Other: Halo G6 e-cigarette

INTERVENTIONS:
Drug: Zonisamide — Zonisamide (100 mg/daily) for 12 weeks.
  Other Names: zonegran
Drug: Bupropion — Extended-release bupropion dosing (150 mg each morning days 1-3, then 300 mg/daily) for the remainder of the 12 weeks.
  Other Names: wellbutrin; Zyban
Other: Halo G6 e-cigarette — G6 e-cigarette for ad libitum use for two weeks prior to complete switch day.
  Other Names: e-cigarette

SUMMARY:
This single-group, small-scale, open-label study (N= 25 to 50) will evaluate the impact of combination zonisamide and bupropion on the process of switching from combustible cigarettes (CC) to an e-cigarette. There will be a data collection period of at least five days to obtain baseline data on use of combustible cigarettes. Participants enrolled in the study will receive a G6 e-cigarette at V2 for ad libitum use. After the first week of e-cigarette use, (at V3) participants will be given zonisamide (100 mg/daily) and will begin extended-release bupropion dosing (150 mg each morning days 1-3, then 300 mg/daily) in addition to continued use of the G6. At each visit, participants will receive enough zonisamide, bupropion, and Halo G6 cartomizers to last until their next study visit. Halo G6 and combination zonisamide and bupropion use will continue until the participant returns for the End-of-Study visit (V7).

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to read and understand the information provided in the ICF.
2. Is 21 to 65 years of age (inclusive) at screening.
3. Smokes at least 10 commercially available cigarettes per day (no brand restrictions), for the last 12 months.
4. Has an expired air CO reading of at least 10 ppm at screening.
5. Interested in switching to an electronic cigarette.
6. Willing and able to comply with the requirements of the study.
7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. Planned use of an FDA-approved smoking cessation product during the study.
4. High blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
5. Body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2.
6. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
7. Has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
8. Taking antidepressants, psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics) or medications that prolong QTc.
9. Use of any of these products in the past 30 days:

   1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, or opiates);
   2. Experimental (investigational) drugs that are unknown to participant;
   3. Chronic opiate use.
10. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
11. Pregnant or nursing (by self-report) or has a positive pregnancy test.
12. Enrollment requirements met.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled into the study but discontinued prior to taken any study drug.
Period: Enrolled in Study
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
Started | 26
Completed | 24
Not Completed | 2
Period: Treatment Period
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
Started | 24
Completed | 23
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Two participants were enrolled into the study but discontinued prior to taken any study drug so analysis is based on the 24 participants who started the study drug.
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Cigarettes smoked per day (CPD) [Mean (Standard Deviation); unit: Cigs smoked per day] — Population: Two participants were enrolled into the study but discontinued prior to taken any study drug so analysis is based on the 24 participants who started the study drug.
  Cigs smoked per day
    number analyzed (Participants) | 24
    (all) | 21.2 (6.64)
FTND -- The Fagerström Test for Nicotine Dependence Score [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is a six-item questionnaire developed by Karl-Olov Fagerström and is used to determine someone's level of nicotine dependence. The scores obtained on the test allow the classification of nicotine dependence in three different levels: mild (0-3 points), moderate (4-6 points), and severe (7 -10 points). Population: Two participants were enrolled into the study but discontinued prior to taken any study drug so analysis is based on the 24 participants who started the study drug.
  units on a scale
    number analyzed (Participants) | 24
    (all) | 6.1 (1.82)
Expired air carbon monoxide (CO) [Mean (Standard Deviation); unit: ppm] — Population: Two participants were enrolled into the study but discontinued prior to taken any study drug so analysis is based on the 24 participants who started the study drug.
  ppm
    number analyzed (Participants) | 24
    (all) | 26.0 (9.19)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Completely Switched From Combustible Cigarettes to Halo G6 E-Cigarettes
Description: Defined as self-report of no cigarette smoking (not even a puff), confirmed by an expired air CO reading of less than 5 ppm.
Time Frame: Weeks 8-11 post-quit date (weeks 10-13 post baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
Number analyzed (Participants) | 24
Participants | 8

2. Secondary Outcome: Point Abstinence From Combustible Cigarettes
Description: Assessed by self-report utilizing an automated SMS messaging system.
Time Frame: Six months post switch day (approximately 6 months post baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
Number analyzed (Participants) | 24
Participants | 15

3. Secondary Outcome: Change in Rewarding Effects of Smoking Combustible Cigarettes
Description: Characterize changes in the two primary scales of the Cigarette Evaluation Questionnaire (mCEQ), assessing smoking satisfaction and psychological reward, compared between cigarettes smoked after meals versus all others smoked during the day, examining how this difference changes after zonisamide/bupropion usage. The mCEQ uses a 7-point scale (0=Not at all; 1=Very little; 2=A little; 3=Moderately; 4=A lot, 5=Quite a lot; 6=Extremely) to measure the following subscales: Satisfaction, Psychological Reward, Enjoyment of Respiratory Tract Sensations, Craving Reduction, Aversion.
Time Frame: First week compared to after start of study drugs (Weeks 2-13 post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
Number analyzed (Participants) | 24
score on a scale
  CEQ Satisfaction Scale | 0 (1.2)
  CEQ Psych Reward Scale | 0.2 (1.1)

ADVERSE EVENTS:
Time Frame: During 13 week study period.
Arm/Group | Combination Zonisamide and Bupropion With E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Zonisamide and Bupropion With E-cigarette (N=24)
Constipation (Gastrointestinal disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (5)
Throat irritation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tinnitus (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Aversion to cigarettes (Nervous system disorders) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2)
Elevated blood pressure (Cardiac disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT04388319/Prot_SAP_000.pdf